CLINICAL TRIAL: NCT03890913
Title: Painted Playgrounds: A Scalable Approach to Increasing Physical Activity and Motor Skills in Louisiana Preschool Aged Children. Aim 1: Observation
Brief Title: Painted Playgrounds Aim 1
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Blue Cross Blue Shield (Other)
Responsible Party: Principal Investigator, Amanda Staiano, Principle Investigator, Pennington Biomedical Research Center
Other Study IDs: PBRC 2017-034
Record Dates: First submitted 2019-01-29; First posted 2019-03-26 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation: All childcare centers enrolled to Aim 1 will be observed. The physical activity environment will be examined before and after the implementation of playground stencils.

SUMMARY:
Painted Playgrounds Aim 1: Observation will examine the physical environment of licensed childcare centers before and after painting stencil activities (hopscotch, foursquare, fun trails, etc.) on playgrounds. The stencils are a promising intervention to help decrease obesity and sedentary behaviors in preschool aged children because they are cost-effective and easily scalable. Observations will be held at follow-ups by video recording during recess and using a modified behavioral observation method, called SOPLAY. Surveys will be administered to childcare center directors to report further on their physical activity environment and how much they are interacting with the stencils.

DETAILED DESCRIPTION:
Preschool is a critical period during which children develop fundamental motor skills, build confidence in their movement, and start a physical activity trajectory that follows through adolescence and beyond. Unfortunately, few sustainable interventions have succeeded in increasing preschool children's physical activity, and subsequently children are developing obesity at alarming rates. A simple, low-cost strategy is the addition of colorful markings (i.e. hopscotch, foursquare, fun trails) to existing playgrounds or open spaces. These "painted playgrounds" have been shown to be effective to increase physical activity in older school-aged children but remain understudied in preschool children. The proposed project will examine the physical activity environment of licensed childcare centers before and after the implementation of a promising (cost-effective, easily scalable) playground stenciling intervention.

The project aim will be achieved through a prospective observational epidemiological approach before and after a stenciling intervention is implemented. Among 4 childcare centers licensed in East Baton Rouge Parish (EBR), the investigators will first observe the playground environment to assess the equipment, space, ground material, etc. to provide a baseline measure of the physical activity environment prior to stenciling and ensure that intervention and control centers have similar playground environments. A modified behavioral observation method, the System for Observing Play and Leisure Activity in Youth (SOPLAY), will be used during recess to identify changes in physical activity after the stencils are added and which stencils are generating the biggest changes in physical activity. Surveys will be administered to center directors to further understand the physical activity environment (i.e. policies, additional PA support, etc.) in each center. This project will examine how a promising (cost-effective, easily scalable) playground stenciling intervention changes the physical activity landscape of childcare centers in order to provide evidence for the need for dissemination to numerous childcare centers across Louisiana. Ultimately, this pilot may launch an innovative strategy that has the potential to disrupt negative trends in obesity and sedentary behavior among Louisiana preschoolers.

ELIGIBILITY:
Inclusion Criteria:

* Licensed by DOE as a Class A or Class B childcare center
* Current childcare enrollment of at least 20 children between the ages of 3-6 years
* Has a playground/play area with adequate space for stenciling

Exclusion Criteria:

* Childcare center and/or childcare center director are unwilling to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Four licensed DOE Class A or B childcare centers will be selected from a list of all DOE licensed childcare centers in East Baton Rouge Parish.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Staiano, PhD, Principal Investigator — Pennington Biomedical
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Webster EK, Kepper MM, Saha S, Beyl RA, Kracht CL, Romain JS, Staiano AE. Painted playgrounds for preschoolers' physical activity and fundamental motor skill improvement: a randomized controlled pilot trial of effectiveness. BMC Pediatr. 2023 Sep 9;23(1):455. doi: 10.1186/s12887-023-04260-2. PMID 37689622

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Childcare Centers
Groups:
- Intervention Centers: All childcare centers enrolled to Aim 1 will be observed. The physical activity environment will be examined before and after the implementation of playground stencils; wait-list control DID have spray painted stencils. 51 preschoolers at 4 childcare centers were observed
- Wait-List Control: All childcare centers enrolled to Aim 1 will be observed. The physical activity environment will be examined before and after the implementation of playground stencils; wait-list control did NOT have spray painted stencils. 51 preschoolers at 4 childcare centers were observed
Period: Overall Study
Arm/Group | Intervention Centers | Wait-List Control
Started | 32; 2 Childcare Centers | 19; 2 Childcare Centers
Completed | 32; 2 Childcare Centers | 19; 2 Childcare Centers
Not Completed | 0; 0 Childcare Centers | 0; 0 Childcare Centers

BASELINE CHARACTERISTICS:
Groups:
- Children Enrolled in Participating Child Care Centers - Control: All childcare centers enrolled to Aim 1 will be observed. The physical activity environment will be examined before and after the implementation of playground stencils; control group DID receive stencils. The demographic data listed represents the 19 children in the control group
- Children Enrolled in Participating Child Care Centers - Intervention: All childcare centers enrolled to Aim 1 will be observed. The physical activity environment will be examined before and after the implementation of playground stencils; intervention group did NOT receive stencils. The demographic data listed represents the 32 children in the intervention group
- Total: Total of all reporting groups
Arm/Group | Children Enrolled in Participating Child Care Centers - Control | Children Enrolled in Participating Child Care Centers - Intervention | Total
Number analyzed (Participants) | 19 | 32 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19 | 32 | 51
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 17 | 29
  Male | 7 | 15 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 23 | 35
  White | 6 | 7 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Children's Physical Activity Levels During Recess
Description: The investigators will observe the number of children participating in physical activity during recess before and after the implementation of a playground stenciling intervention to asses for change. The observation will be performed using a modified version of the System for Observing Play and Leisure Activity in Youth (SOPLAY). SOPLAY is an observational tool designed to assess physical activity levels & environmental conditions in settings where youth are engaged in play and leisure. SOPLAY is typically used to capture data on physical activity levels, the type of activity, and environmental factors that may influence youth activity. SOPLAY does not produce a single cumulative "score" but instead provides a detailed record of activity levels and environmental conditions. The data is typically analyzed to assess patterns, identify factors that promote or inhibit physical activity, and guide interventions to improve youth physical activity engagement.
Time Frame: Children will be examined at follow up (6-8 weeks after receiving the stencils)
Population: A total number of 45 children were observed playing in either the intervention or control playgrounds. When the numbers listed below does not match with the over number of participants analyzed (51), that means the children not represented DID NOT use the stencils at their center. Reminder that the participants listed below are children who were students at the 4 sites within this aim.
Measure: Mean (Standard Deviation); unit: count of participants
Groups:
- Children Enrolled in Participating Child Care Centers - Control: All childcare centers & the children within that center enrolled to Aim 1 will be observed. The physical activity environment will be examined before and after the implementation of playground stencils; control group DID receive stencils. The demographic data listed represents the 19 children in the control group
- Children Enrolled in Participating Child Care Centers - Intervention: All childcare centers & the children within that center enrolled to Aim 1 will be observed. The physical activity environment will be examined before and after the implementation of playground stencils; intervention group did NOT receive stencils. The demographic data listed represents the 32 children in the intervention group
Arm/Group | Children Enrolled in Participating Child Care Centers - Control | Children Enrolled in Participating Child Care Centers - Intervention
Number analyzed (Participants) | 19 | 26
count of participants
  Light physical activity | 2.3 (3.3) | 4.3 (2.9)
  Moderate physical activity | 3.5 (3.6) | 0.5 (3.2)
  Vigorous PA | 2.6 (1.2) | .9 (1.1)
  Moderate-to-Vigorous Physical Activity | 6.2 (4.1) | 1.4 (3.7)
  Sedentary Behavior | -8.5 (6.8) | -5.6 (6.1)

2. Secondary Outcome: Childcare Center Physical Activity Environment
Description: Childcare center directors will complete a survey assessing the physical activity environment (e.g. policies for outdoor play and screen time, available equipment, teacher engagement in physical activity, etc.) of their childcare center.
Time Frame: Baseline
Population: 4 sites were selected to participate in this study thus 4 directors completed the survey for this aim; directors were not considered to be enrolled in the study. These 4 centers are where the 51 preschoolers attend school and where the stencils were painted; child participants were not included in this analysis.
Measure: Count of Units; unit: childcare centers
Units Other Than Participants: childcare centers
Groups:
- Observation: All childcare centers enrolled to Aim 1 will be observed. The physical activity environment will be examined before and after the implementation of playground stencils. 51 preschoolers at 4 childcare centers were observed
Arm/Group | Observation
Number analyzed (Participants) | NA
Number analyzed (childcare centers) | 4
childcare centers
  Does your center offered structured programs children to be physically active?: Yes | 2
  Does your center offered structured programs children to be physically active?: No | 2
  Do any community organizations support or provide physical activity programs at the center?: Yes | 3
  Do any community organizations support or provide physical activity programs at the center?: No | 1
  Active play time is provided to all preschool children more than 120 minutes each day.: Yes | 4
  Active play time is provided to all preschool children more than 120 minutes each day.: No | 0
  Preschool children are expected to remain seated for no more than 15 minutes at a time.: Yes | 2
  Preschool children are expected to remain seated for no more than 15 minutes at a time.: No | 2
  Indoor gross motor play area for preschool children consists of space for all activities.: Yes | 1
  Indoor gross motor play area for preschool children consists of space for all activities.: No | 3
  Outdoor play areas consist of multiple play areas, open space, and a track/path for wheeled toys.: Yes | 4
  Outdoor play areas consist of multiple play areas, open space, and a track/path for wheeled toys.: No | 0
  Portable play equipment consists of lots of variety for children to use at the same time.: Yes | 1
  Portable play equipment consists of lots of variety for children to use at the same time.: No | 3
  Providers are offered training opportunities in physical activity at 2 or more times per year.: Yes | 2
  Providers are offered training opportunities in physical activity at 2 or more times per year.: No | 2

3. Secondary Outcome: Satisfaction With Playground Stencils
Description: Intervention Childcare center directors will complete a survey to measure their satisfaction and perceptions of teacher's satisfaction with the playground stencils.
Time Frame: 6-8 weeks after receiving the playground stencils.
Population: 4 sites were selected to participate in this study; 2 were in the intervention group & 2 were in the control group. These 4 centers are where the 51 preschoolers attend school and where the stencils were painted. The 2 directors from the intervention group only are included in the analysis population.
Measure: Count of Units; unit: childcare centers
Units Other Than Participants: childcare centers
Groups:
- Observation: Childcare centers enrolled in the intervention group of Aim 1 will be observed. The physical activity environment will be examined before and after the implementation of playground stencils.
Arm/Group | Observation
Number analyzed (Participants) | 2
Number analyzed (childcare centers) | 2
childcare centers
  Do providers use the playground to teach academic concepts through movement?: Yes | 2
  Do providers use the playground to teach academic concepts through movement?: No | 0
  If yes, are stencils used?: Yes | 1
  If yes, are stencils used?: No | 1
  Have you seen any change in students' physical activity since the playground stencils were painted?: Yes | 1
  Have you seen any change in students' physical activity since the playground stencils were painted?: No | 1
  Are playground stencils used to infuse physical activity into the day outside of recess?: Yes | 0
  Are playground stencils used to infuse physical activity into the day outside of recess?: No | 2

4. Secondary Outcome: Childcare Center Resources for Physical Activity
Description: Project staff will evaluate the availability of resources (i.e. playground space, equipment, etc.) at each childcare center.
Time Frame: Baseline
Population: as for outcome 3
Measure: Count of Units; unit: childcare centers
Units Other Than Participants: childcare centers
Arm/Group | Observation
Number analyzed (Participants) | 2
Number analyzed (childcare centers) | 2
childcare centers
  Was Portable Play Equipment Present?: Yes | 1
  Was Portable Play Equipment Present?: No | 1
  Was Fixed Play Equipment Present?: Yes | 2
  Was Fixed Play Equipment Present?: No | 0

ADVERSE EVENTS:
Time Frame: 8 weeks
Groups:
- Children Enrolled in Participating Child Care Centers - Control: All childcare centers enrolled to Aim 1 will be observed. The physical activity environment will be examined before and after the implementation of playground stencils. 19 preschoolers at 4 childcare centers were in the control group.
- Children Enrolled in Participating Child Care Centers - Intervention: All childcare centers enrolled to Aim 1 will be observed. The physical activity environment will be examined before and after the implementation of playground stencils. 32 preschoolers at 4 childcare centers were in the intervention group.
Arm/Group | Children Enrolled in Participating Child Care Centers - Control | Children Enrolled in Participating Child Care Centers - Intervention
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/32
Other Adverse Events (participants affected / at risk) | 0/19 | 0/32

LIMITATIONS AND CAVEATS:
Limitations include the small sample for this pilot study. Only four schools were examined in one region of the United States, so results may only be generalizable to this area or to programs with similar characteristics. The limited access to concrete space in most ECE centers is a limitation that must be considered for the expansion of this intervention. Finally, intervention fidelity was not measured, nor was PA measured immediately after introducing the markings on the playground.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-30): https://cdn.clinicaltrials.gov/large-docs/13/NCT03890913/Prot_SAP_000.pdf